CLINICAL TRIAL: NCT05243056
Title: Piloting Y-AMBIENT: A Quality of Life Intervention for Young African American Breast Cancer Survivors in Treatment
Brief Title: A Quality of Life Intervention for Young African American Breast Cancer Survivors in Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Timiya Nolan, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-300012132; K08CA245208 (NIH); NCI-2021-02286 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-11-10; First posted 2022-02-16 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-05

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (Y-AMBIENT) (Experimental): Patients receive three themed education sessions over 1 hour each, written materials, and videos at month 1. Patients also participate in 3, 20 minutes telephone reinforcement calls to discuss how they are doing and discuss any concerns that they are still managing at months 2, 3, and 4.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (enhanced usual care) (Active Comparator): Patients receive usual care at month 1. Patients also participate in 3, 20 minutes telephone reinforcement calls to discuss their chemotherapy regimen at months 2, 3, and 4.
  Interventions: Other: Best Practice; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive enhanced usual care
  Other Names: standard of care; standard therapy
  Arms: Arm II (enhanced usual care)
Other: Educational Intervention — Receive Y-AMBIENT
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Arm I (Y-AMBIENT)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the use of a quality of life intervention called Y-AMBIENT to help young African American with stage I-III breast cancer manage daily life. Y-AMBIENT is a four-month, telephone-based intervention that includes three themed education sessions with three follow-up sessions, written materials, and videos. The Y-AMBIENT intervention may improve quality of life and other health-related outcomes in young African American breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate feasibility and acceptability of Y-AMBIENT and enhanced usual care among young African American breast cancer survivors.

II. Explore the degree to which the Y-AMBIENT versus (vs.) enhanced usual care affects preliminary health-related outcomes among young African American (AA survivors).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (Y-AMBIENT): Patients receive three themed education sessions over 1 hour each, written materials, and videos at month 1. Patients also participate in 3, 20 minutes telephone reinforcement calls to discuss how they are doing and discuss any concerns that they are still managing at months 2, 3, and 4.

ARM II (ENHANCED USUAL CARE): Patients receive usual care at month 1. Patients also participate in 3, 20 minutes telephone reinforcement calls to discuss their chemotherapy regimen at months 2, 3, and 4.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Biologically born women
* Self-identify as AA
* Are aged 18 to 44 years on study entry
* Are diagnosed with breast cancer stage I-III
* Are in treatment with chemotherapy and/or radiation for stage I-III breast cancer at study entry
* Are English- speaking
* Have telephone and internet access

Exclusion Criteria:

* Participation in formal survivorship navigation programs because they are associated with improved health- related outcomes, which could be a confounder

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of screen-eligible patients enrolled by consent | Up to 2 years
  Descriptive statistics will be used to compute the proportion of screen-eligible patients enrolled by consent. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Proportion of patients that complete all (seven) study contacts of intervention | Up to 2 years
  Descriptive statistics will be used to compute proportion of patients that complete all (seven) study contacts of the intervention. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Acceptability/Relevance of Intervention Sessions | Up to 2 years
  Will use qualitative interview to assess participants' perceptions of its acceptability/relevance of each of the six study contacts, using a Likert scale 0 to 10 with 0 being not at all satisfied/useful and 10 being completely satisfied/useful and an open ended question to understand why each score was provided. A composite score will be determined, where higher scores equate to higher acceptability/relevance. Descriptive statistics will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate. Qualitative responses will be analyzed for content.
Participation in aspects of protocol | Up to 2 years
  Will use qualitative interview to assess participants' engagement by review of task completion to participate in aspects of the protocol (as an indicator of participant burden). There are a total of six sessions to complete and seven videos to review. Descriptive statistics will be used to compute the proportion of participant self-reported effectiveness of each intervention via the logs. Completion of tasks indicates greater willingness to participate.
Use of proposed self-management strategies and perceived effectiveness | Up to 2 years
  Will use qualitative interview to assess participants' engagement by review of use of proposed self-management strategies and their perceived effect on quality of life concerns using a Likert scale 0 to 10 with 0 being not at all effective and 10 being most effective. Descriptive statistics will be used to compute the proportion of participant self-reported effectiveness of each intervention via the logs. Qualitative responses will be analyzed for content.
Medical Outcomes Survey Short-Form (SF-36) | Baseline up to 1 month post-intervention
  The SF-36 is a well-established measure of health status in cancer survivors. SF-36 includes one multi-item scale assessing eight health concepts: limitations in physical activity, social activity, role activity, bodily pain, psychological distress, limitations in social activity due to emotional distress, vitality, and general health perceptions. The scale ranges from 0-100. Higher scores indicate better functioning.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
PROMIS Global Health10 | Baseline up to 1 month post-intervention
  The PROMIS Global Health 10 is a well-established measure of health status in cancer survivors. It assesses health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. Higher scores indicate better functioning.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
(Functional Assessment of Chronic Illness Therapy Spiritual Well-Being (FACT-Sp 12) | Baseline up to 1 month post-intervention
  The FACIT-SP-12 is the most widely used measure of spiritual well-being among those with cancer. Its subscales measure faith, meaning, and peace. Higher scores reflect higher well-being.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
MOS Modified Social Support Survey | Baseline up to 1 month post-intervention
  MOS assesses dimensions of social support with four functional support scales: emotional/informational, tangible, affectionate, and positive social interaction. The scale ranges from 0-100. Higher scores indicate greater social support.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
COmprehensive Score for Financial Toxicity [COST]-Functional Assessment of Chronic Illness Therapy [FACIT] | Baseline up to 1 month post-intervention
  COST-FACIT is a measure of financial toxicity and/or concerns related to cost of cancer care. Lower COST scores indicate higher financial toxicity.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
PROMIS Applied Cognition - General Concerns short form (8- item) | Baseline up to 1 month post-intervention
  This instrument measures working memory, speed of processing, and executive control of cognitive functioning. Higher scores reflect higher perceived cognitive functionality.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
Perceived Stress | Baseline up to 1 month post-intervention
  This instrument measures the perception of stress.
  The PSS was designed for use in community samples with at least a junior high school education. The items are easy to understand, and the response alternatives are simple to grasp. This study will be using a short scale version of the scale, which uses four of the questions (2,4,5, and 10) of the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Timiya Nolan, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu